CLINICAL TRIAL: NCT07190495
Title: Preoperative Ginger for the Prevention of Postoperative Nausea and Vomiting in Patients Undergoing Laparoscopic Cholecystectomy: A Double-Blind Randomized Controlled Trial
Brief Title: Ginger to Prevent Nausea and Vomiting After Laparoscopic Cholecystectomy
Acronym: GINGER-PONV
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Ben Taleb Ibtissem, Assistant Professor in Anesthesiology and Intensive Care, University Tunis El Manar
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GINGER PONV
Record Dates: First submitted 2025-09-14; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Postoperative Nausea and Vomiting; Laparoscopic Cholecystectomy
Keywords: Ginger; Postoperative Nausea and Vomiting; Laparoscopic Cholecystectomy
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — ginger extract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ginger group (Active Comparator): Patients will receive 800 mg of oral ginger 2 hours before laparoscopic cholecystectomy
  Interventions: Drug: Ginger
- Placebo group (Placebo Comparator): Patients will receive an oral placebo capsule identical in appearance to ginger, administered 2 hours before laparoscopic cholecystectomy
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ginger — Patients will receive 800 mg of oral ginger 2 hours before laparoscopic cholecystectomy
  Arms: Ginger group
Drug: Placebo — Patients will receive an oral placebo capsule identical in appearance to ginger, administered 2 hours before laparoscopic cholecystectomy
  Arms: Placebo group

SUMMARY:
This study aims to evaluate whether preoperative oral administration of ginger (800 mg, given 2 hours before surgery) reduces the incidence and severity of postoperative nausea and vomiting (PONV) within the first 24 hours after laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Scheduled for elective laparoscopic cholecystectomy under general anesthesia.
* American Society of Anesthesiologists (ASA) physical status I-III.
* Able to understand the study procedures and provide written informed consent.

Exclusion Criteria:

* Known allergy or hypersensitivity to ginger
* Documented history of bleeding disorders or current treatment with anticoagulant agents
* History of severe postoperative nausea and vomiting or an Apfel score of 4
* Administration of antiemetic drugs or corticosteroids during the preoperative period
* Pregnancy or breastfeeding
* Active gastrointestinal or liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-07-05 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative nausea and vomiting (PONV) within 2 hours post-surgery | 2 hours after surgery.
  Occurrence of at least one episode of nausea or vomiting within the first 2 hours after surgery.

SECONDARY OUTCOMES:
Recurrence of PONV beyond 2 hours postoperatively | From 2 hours to 24 hours after surgery.
  Proportion of participants who experienced at least one additional episode of nausea or vomiting occurring after the 2-hour postoperative time point.
Incidence of postoperative nausea and vomiting (PONV) within 24 hours post-surgery | 24 hours after surgery.
  Occurrence of at least one episode of nausea or vomiting within the first 24 hours after surgery.
Total number of vomiting episodes | Within 24 hours post-surgery.
  Cumulative number of vomiting episodes recorded per participant during the first 24 hours after surgery.
Use of rescue antiemetics | 24 hours postoperatively
  The need for rescue antiemetics within 24 hours postoperatively.
Incidence of ginger-related adverse events | Within 24 hours after surgery
  Number of participants experiencing adverse events known to be associated with ginger, including gastrointestinal discomfort (heartburn, abdominal pain, bloating, diarrhea), bleeding, or allergic reactions in the 24 hours after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamed Taher Maamouri University Hospital, Nabeul, Nabeul Governorate, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided